CLINICAL TRIAL: NCT04181359
Title: The Effect of Inhaled Nitric Oxide on Dyspnea and Exercise Tolerance in Interstitial Lung Disease.
Acronym: iNO
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was no longer feasible as designed.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00092702
Record Dates: First submitted 2019-11-21; First posted 2019-11-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide (Experimental): Inhaled nitric oxide, which consists of breathing medical grade air (21% O2) with 40 parts per million of nitric oxide.
  Interventions: Drug: Nitric Oxide
- Placebo (Placebo Comparator): Inhaled placebo, which consists of breathing medical grade air (21% O2).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitric Oxide — Inhaled nitric oxide, which consists of breathing medical grade air (21% O2) with 40 parts per million of nitric oxide.
  Other Names: iNO
  Arms: Nitric Oxide
Drug: Placebo — Inhaled placebo, which consists of breathing medical grade air (21% O2).
  Arms: Placebo

SUMMARY:
Interstitial Lung Disease (ILD) is a is a lung disorder which makes breathing more difficult. During exercise, patients with ILD are not efficient breathers and this leads to serious breathing difficulties, which often causes these patients to stop exercise at low intensities. The investigators think that these patients with ILD have problems exchanging fresh gas (i.e., oxygen) into the blood stream because of poor lung blood vessel function. The investigators will test whether inhaled medications, specifically nitric oxide, can improve lung blood vessel function and decrease breathing difficulties during exercise. With this research, the investigators will understand more about breathing efficiency and lung blood vessel function in mild ILD patients, and find out whether improving lung blood vessel function helps ILD patients breathe easier and exercise longer. Understanding the reasons behind the feeling of difficult breathing may lead to more effective therapy and improved quality of life in ILD patients.

DETAILED DESCRIPTION:
BACKGROUND

Interstitial Lung Disease (ILD) is a respiratory disorder characterized by chronic inflammation and fibrosis of the lung parenchyma. Exertional dyspnea (perceived breathlessness) is a hallmark of ILD regardless of severity and is the primary reason for the observed exercise intolerance, typically observed in this population. Dyspnea in ILD has been shown to profoundly reduce quality of life, physical activity, and impair the ability of participants with ILD to complete day-to-day tasks. Previous work in ILD has demonstrated that exertional dyspnea is the result of increased work of breathing during exercise, and that this increased work of breathing comes from: 1) an exaggerated ventilatory response to exercise (i.e. increased minute ventilation relative to carbon dioxide production, V̇E/V̇CO2), and 2) airflow limitation (i.e. expiratory flow limitation and resulting dynamic hyperinflation). A growing body of work has focused on respiratory mechanics in ILD; however, very little has been done to understand and treat the exaggerated ventilatory response to exercise in ILD.

Several previous studies in ILD have consistently shown an elevated ventilatory response (i.e. greater V̇E/V̇CO2) during exercise. This increased V̇E/V̇CO2 in ILD appears to be secondary to increased deadspace ventilation (i.e. sections of the lung with ventilation, but no perfusion), and this increased deadspace ventilation results in a compensatory increase in total minute ventilation (i.e. increased V̇E/V̇CO2) to maintain effective alveolar ventilation and arterial blood gas homeostasis. The underlying mechanism(s) for the increased deadspace ventilation and V̇E/V̇CO2 during exercise in mild ILD is currently unclear; however, pulmonary microvascular abnormalities and hypoperfusion of pulmonary capillaries are potential pathophysiologic mechanisms. Individuals with ILD have a reduced pulmonary capillary blood volume and, in more severe ILD, present with pulmonary vascular dysfunction and are prone to developing exercise-induced pulmonary arterial hypertension. It is likely that the pulmonary vascular dysfunction, in ILD, may impair pulmonary capillary perfusion, leading to ventilation (V̇A) -perfusion (Q̇) inequality (specifically, areas of high, V̇A/Q̇, which is indicative of increased deadspace), however this has not yet been examined. Inhaled nitric oxide (NO) is commonly used to test for pulmonary vasodilatory responses in individuals with pulmonary arterial hypertension (PAH), as it increases NO bioavailability and improves pulmonary vascular function. Previous work in PAH and heart failure (HF) has shown that standard doses (20-40 parts per million (ppm)) of inhaled NO can reduce pulmonary vascular resistance and increase peak oxygen consumption (V̇O2peak). If inhaled NO can reduce vascular dysfunction and increase perfusion in ILD, this would result in a reduction in V̇E/V̇CO2 and dyspnea, and improved exercise tolerance.

STUDY PURPOSE

Purpose: To examine the effect of inhaled NO on exercise capacity (V̇O2peak), ventilation and dyspnea in ILD.

Hypothesis: Inhaled NO will improve exercise capacity, secondary to reduced V̇E/V̇CO2 and dyspnea, in individuals with ILD.

Study Design: Randomized double-blind cross-over design.

Study Protocol:

Six sessions will be completed over a 3-week period in the following order: Day 1) Participant enrollment, medical history, standard pulmonary function (PFT) and cardiopulmonary exercise test (CPET). Days 2 & 3) Randomly-ordered experimental CPETs while either breathing room air or inhaled nitric oxide (room air with 40 ppm NO). Days 4 & 5) Randomly-ordered constant load exercise tests, at 75% peak power output, while either breathing room air or inhaled nitric oxide (room air with 40 ppm NO). Day 6) Resting and exercise trials while breathing room air or inhaled nitric oxide with ultrasonography doppler measurements to determine pulmonary arterial systolic pressure. Each visit will take approximately 3 hours.

On Day 1, participants will complete the informed consent procedure, fill out a medical history questionnaire and be screened for exercise using the physical activity readiness questionnaire. Study participants will undergo lung function and cardiopulmonary exercise testing on the same day. The participants will be spending approximately three hours in the laboratory on this testing day.

On days 2 & 3 (one day per week in 2 consecutive weeks; order randomized), the participants will breathe the placebo, which is medical grade air (room air) or room air titrated with 40 parts per million of nitric oxide and have blood flow/cardiac output and expired gas evaluated, and time to exhaustion determined in a standard incremental cardiopulmonary exercise test.

On day 2, the participant will lie supine and be rested for 5 minutes. Resting blood pressure will be determined using manual auscultation. Resting cardiac output will be evaluated using noninvasive impedance cardiography (PhysioflowTM) and oxygen saturation estimated with pulse oximetry. Ventilation will be measured from expired gas analysis. Following these measurements, the subject will begin to breathe medical grade room air. Following a 20 minute wash-in period, ventilation, cardiac output and oxygen saturation recordings will be repeated. Participants will then perform a standard cardiopulmonary exercise test while continuing to breathe the medical grade room air. The participants will be spending approximately three hours in the laboratory on this testing day.

Day 3 will be identical to day 2 except, in the place of medical grade room air, participants will breathe room air with 40 parts per million of nitric oxide.

On days 4 & 5 (one day per week in 2 consecutive weeks; order randomized), the participants will breathe the placebo, which is medical grade air (room air) or room air titrated with 40 parts per million of nitric oxide and have blood flow/cardiac output and expired gas evaluated, and time to exhaustion determined in a standard constant work rate cardiopulmonary exercise test. Measurement procedures will be identical to days 2 & 3.

On day 6, the participants will complete resting and sub-maximal exercise trials while breathing placebo or iNO, with ultrasonography Doppler measurements to determine pulmonary arterial systolic pressure.

The participant will lie supine and be rested for 5 minutes. Resting blood pressure will be determined using manual auscultation and pulmonary arterial pressure by echocardiography. Resting cardiac output will be evaluated using impedance cardiography (PhysioflowTM) and oxygen saturation estimated with pulse oximetry. Ventilation will be measured from expired gas analysis. Following these measurements, the subject will begin to breathe either placebo or iNO. Upon completion of resting measurements, participants will complete 5-minutes of sub-maximal exercise at 40 Watts in each experimental conditions. All resting measurements will be repeated during exercise. At least 10-minute recover will be given between conditions to ensure washout of NO and restoration of baseline oxygen saturation.

Intervention

Inhaled Nitric Oxide Intervention: Inhaled NO is a selective pulmonary vasodilator and has been shown to improve blood flow to well-ventilated lung areas (i.e. improve V̇A/Q̇ matching) in conditions with elevated vascular tone. Inhaled NO has been previously shown to lower pulmonary artery pressure during exercise in individuals with severe lung disease, while not affecting systemic blood pressure. It is important to note that a selective pulmonary vasodilator will be used instead of an intravenously infused vasodilator (e.g. prostacyclin) to avoid systemic vasodilation, severe arterial hypotension and syncope. Consistent with previous work, a standard 40 ppm dose of inhaled NO will be administered using a non-rebreathing circuit.

Statistical analysis and Interpretation: A 2-way repeated measures ANOVA will be used to evaluate the changes in V̇E/V̇CO2, dyspnea and exercise capacity (V̇O2peak) with inhaled NO during exercise. Type of intervention (room air vs inhaled NO), and time-point (baseline and during exercise) will be used as fixed factors in the statistical analysis. Should inhaled NO reduce V̇E/V̇CO2 and dyspnea, and improve exercise capacity in ILD, these results would indicate that pulmonary vascular dysfunction contributes to exercise intolerance as well as the potentiated ventilatory and dyspnea response to exercise in participants with ILD.

ELIGIBILITY:
Inclusion Criteria:

* ILD participants free of any significant cardiovascular, metabolic or neuromuscular disease. Specific criteria are:
* Established physician diagnosis of ILD
* Forced vital capacity 50-80 % predicted
* Diffusing capacity for carbon monoxide 35-60 % predicted
* Able to complete a 6-minute walk test
* Participants will range from 18-85 years old.
* There are no restrictions on pulmonary medications, however, participants will be asked to withdraw from long-acting beta agonists 48 hours prior to trials.

Exclusion Criteria:

* Participants with current or previous history of myocardial infarction or angina pectoris will be excluded.
* Participants with a lowest arterial oxygen saturation < 84% during the initial CPET (day 1) on room air will be excluded.
* Patient receiving treatment for isosorbide mononitrate or pulmonary arterial hypertension (PAH) medications will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | Within 20-25 minutes post-dose
  Exercise capacity as determined by peak power output and oxygen uptake (V̇O2peak).

SECONDARY OUTCOMES:
Ventilation | Within 20-25 minutes post-dose
  Ventilatory responses during exercise (i.e. V̇E/V̇CO2)
Perceived breathing discomfort (Modified Borg 0-10 categorical ratio scale) | Within 20-25 minutes post-dose
  Perceived breathing discomfort during exercise, also termed exertional dyspnea. Participants will rate their perceived breathing discomfort on a modified Borg categorical ratio scale (0-10). 0 indicates no breathing discomfort and 10 indicates maximal breathing discomfort.
Pulmonary vascular function | Within 5 minutes post-dose
  Pulmonary artery systolic pressure at rest

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ferrara, MD, Principal Investigator — University of Alberta; Michael Stickland, PhD, Study Director — University of Alberta

IPD SHARING:
Plan to Share IPD: No